CLINICAL TRIAL: NCT00628979
Title: Addressing Help-Seeking Barriers in Developing an Intensive Treatment for Veterans With Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Teng, Ellen - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRECC004
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): CBT
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — cognitive- behavioral treatment for panic disorder.

SUMMARY:
The purpose of this study is to understand some of the reasons why recently deployed veterans decline psychosocial treatment options for panic disorder and to test a brief weekend treatment for panic attacks.

DETAILED DESCRIPTION:
The population of interest for this program includes men and women returning from deployment in Iraq or Afghanistan who are seen in the TRP at the MEDVAMC. The study consists of two parts: PART 1 involves a qualitative investigation of treatment-seeking barriers specific to persons who refuse standard treatments and PART 2 is a pilot intervention to treat panic symptoms in service members who have co-existing PTSD symptoms. PART 1 will include approximately 15 individuals who will be interviewed by a member of the study staff. Patients will be interviewed individually following a semi-structured questionnaire designed to help identify treatment-seeking barriers. PART 2 will include 8 individuals who will be enrolled in an open-trial of a two-day intensive cognitive-behavioral treatment for panic disorder, which will occur over the weekend. No participants will be assigned to a control condition. All activities related to this project including the interviews and intervention will be delivered in either the TRP at the MEDVAMC or at the Houston Center for Quality of Care and Utilization Studies (HCQCUS), a nearby facility.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans;
2. age 18-74;
3. current diagnosis of panic disorder;
4. PTSD symptoms that either meet full diagnostic criteria from the Diagnostic and Statistical Manual-Fourth Edition (DSM-IV) or are at a sub-clinical level. Sub-clinical PTSD is defined as patients who meet either PTSD criteria B and C or B and D, but fail to meet all three;
5. panic disorder and PTSD present for at least 1 month;
6. PART 1 only: patients who are clinically eligible to participate in the study and refuse standard psychosocial treatments (e.g., 12 weeks of cognitive behavioral therapy) for panic disorder.

Exclusion Criteria:

1. Current substance dependence;
2. diagnosed with bipolar disorder or psychosis;
3. current suicidal/homicidal ideation and intent;
4. severe depression (precluding participation in a research study);
5. panic attacks related only to a diagnosis of a specific phobia;
6. medical conditions mimicing anxiety (e.g., mitral valve prolapse);
7. PART 1 only: patients who are clinically eligible for the study and are willing to engage in a minimum of 12 weeks of psychosocial treatment for panic disorder.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Qualitative data regarding treatment seeking barriers | 6 months

SECONDARY OUTCOMES:
Panic attack frequency and severity; treatment acceptability | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Teng, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center (152)
Locations (1):
- Michael E. DeBakey VA Medical Center (152), Houston, Texas, United States